CLINICAL TRIAL: NCT05965466
Title: Effect of Gastric Cancer Surgical Resection Extent on Postoperative Gallstone Formation: A Retrospected Cohort Study
Brief Title: The Incidence of Gallstones After Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGBS
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Gallstone; Gastric Cancer
Keywords: Gallstone; Gastric Cancer; Gastrectomy
MeSH Terms: conditions — Gallstones; Stomach Neoplasms | interventions — Gastroenterostomy

STUDY DESIGN:
Intervention Model Description: Distal gastrectomy and Total gastrectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal gastrectomy (Experimental): Distal subtotal gastrectomy was performed after exclusion of contraindications to surgery. Gastrointestinal reconstruction was performed by residual gastrojejunal Roux-en-Y anastomosis. Anastomosis was performed ex vivo or in vivo.
  Interventions: Procedure: Distal gastrectomy and radical resection
- Total gastrectomy (Sham Comparator): Total gastrectomy was performed after the exclusion of contraindications to surgery. Gastrointestinal reconstruction was performed by oesophageal jejunum Roux-en-Y anastomosis. Anastomosis was performed ex vivo or in vivo.
  Interventions: Procedure: Total gastrectomy and radical resection

INTERVENTIONS:
Procedure: Distal gastrectomy and radical resection — Distal gastrectomy and Roux-en-Y anastomosis
  Arms: Distal gastrectomy
Procedure: Total gastrectomy and radical resection — Total gastrectomy and Roux-en-Y anastomosis
  Arms: Total gastrectomy

SUMMARY:
To provide preventive and therapeutic strategies for participants with gallstones after gastric cancer by comparing the risk of postoperative gallbladder stone formation with two different resection ranges using the Roux-en-Y reconstruction modality in radical gastric cancer surgery.

DETAILED DESCRIPTION:
A large number of clinical studies have found that the incidence of gallstones in patients after radical gastric cancer surgery is higher than that in the normal population. However, the pathogenesis has not been clarified, and the prophylactic removal of the gallbladder in patients with gastric cancer remains controversial. A previous study found a statistically significant incidence of gallbladder stones after Billroth I versus Roux-en-Y in distal gastrectomy for gastric cancer. Therefore, the investigators plan to conduct a retrospected cohort study to collect further participants with gastric cancer who underwent total gastrectomy to answer whether different surgical resection ranges during surgery increase the incidence of gallstones this question.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Gastric Cancer underwent Gastrectomy

Exclusion Criteria:

* Age less than 18 years or age greater than 75 years;
* Not Roux-en-Y reconstruction;
* R0 excision is not achieved;
* Previous history of upper abdominal surgery, such as cholecystectomy, gastrectomy;
* Preoperative gallbladder diseases, such as gallstones, gallbladder polyps, chronic cholecystitis;
* Preoperative neoadjuvant chemotherapy or radiotherapy;
* Previous history of malignant tumours;
* Patients with mental or developmental abnormalities or women during pregnancy or breastfeeding;
* Gastric perforation or bleeding leading to emergency surgery;
* Palliative surgical treatment;
* Incomplete case information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
Number of gallstone patients | 5years
  Two groups of patients with gastric cancer had a follow-up for more than one year and the number of patients with gallbladder stones on B-ultrasound or Computed Tomography (CT)

SECONDARY OUTCOMES:
Number of patients with postoperative complications | 5years
  The number of patients with postoperative complications such as abdominal haemorrhage, fistula, nausea, vomiting, abdominal infection and incision infection in 2 groups of gastric cancer patients
Number of patients with bile duct stones | 5years
  Two groups of patients with gastric cancer had a follow-up for more than one year. Clinical signs such as Charcot's triad and ultrasound, Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) show the number of patients with bile duct stones

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (2):
- China (2):
  - Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu
  - Wuwei Tumor Hospital, Wuwei, Gansu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park DJ, Kim KH, Park YS, Ahn SH, Park do J, Kim HH. Risk Factors for Gallstone Formation after Surgery for Gastric Cancer. J Gastric Cancer. 2016 Jun;16(2):98-104. doi: 10.5230/jgc.2016.16.2.98. Epub 2016 Jun 24. PMID 27433395
- [Result] Wu CH, Huang KH, Chen MH, Fang WL, Chao Y, Lo SS, Li AF, Wu CW, Shyr YM. Comparison of the Long-term Outcome Between Billroth-I and Roux-en-Y Reconstruction Following Distal Gastrectomy for Gastric Cancer. J Gastrointest Surg. 2021 Aug;25(8):1955-1961. doi: 10.1007/s11605-020-04867-1. Epub 2020 Nov 17. PMID 33205309
- [Derived] Zhang B, Nie P, Lin Y, Ma Z, Ma G, Wang Y, Ma Y, Zhao J, Zhang J, Yue P, Jiang N, Zhang X, Tian L, Lu L, Yuan J, Meng W. High incidence of gallstones after Roux-en-Y reconstruction gastrectomy in gastric cancer: a multicenter, long-term cohort study. Int J Surg. 2024 Apr 1;110(4):2253-2262. doi: 10.1097/JS9.0000000000001136. PMID 38320088